CLINICAL TRIAL: NCT05298761
Title: Efficacy of IV Lignocaine Versus IV Nalbuphine for Attenuation of Pressor Response Diring Laryngoscopy and Intubation in Patients Planned for Thyroid Surgery
Brief Title: Efficacy of I/v Nalbuphine v/s Iv Lignocain in Attanuation of Pressor Responseduring Laryngeoscopy and Intubation in Middle Age Patient Planned for Thyroid Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Amna Sarwar, Principle investigator, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ASarwar
Record Dates: First submitted 2022-02-22; First posted 2022-03-28 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Hemodynamic Stability
MeSH Terms: interventions — Lidocaine; Nalbuphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lignocain (Experimental): I/V lignocain 1.5mg per kg given to participants in state dose
  Interventions: Drug: Lignocaine
- nalbuphine (Experimental): I/v nalbuphine 0.1mg per kg given to participants in stat dose
  Interventions: Drug: Lignocaine

INTERVENTIONS:
Drug: Lignocaine — Inj lignocain and inj nalbuphine given to two groups of participants and effects of both drugs
  Other Names: Nalbuphine

SUMMARY:
Comparison of I/V nalbuphine versus I/V xylocain in attanuation of pressor response during intubation and laryngeoscopy in patients undergoing for thyroid surgery,selection of better supressor agent minimises the drug repated side effects like hypertention tachycardia but also helps in heamodynamically stability at induction.

ELIGIBILITY:
Inclusion Criteria:

* middle age(18_40)
* Asa 1 and 2
* Non hypertensive
* Thyroid patients
* patient who gives consent

Exclusion Criteria:

* hypertensive
* Asa 3 and 4
* Patient refusal

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduce stress response during intubation and hemodynamic stabilty | 10 minutes
  Assesment of Hemodynamic stability by observing vital signs
Achieve hemodynamic stabilty and smooth intubation | 10 minutes
  Assesment of hemodynamic stability by clinical examination of vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Dr.amna Sarwar, Fcps, Principal Investigator — Sheikh zaied medical hospital
Locations (1):
- Dr.amna, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No